CLINICAL TRIAL: NCT03745729
Title: A Single-center, Prospective, Randomized, Double-blind, Controlled Trial for the Effect of Allopurinol Sustained-release Capsules on the Stability of Coronary Plaques in Patients With Acute Coronary Syndrome
Brief Title: Allopurinol in Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Head of department of cardiology, Wuhan Union Hospital, China, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChiCTR1800019389
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: allopurinol sustained-release capsules
- Control group (Placebo Comparator)
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: allopurinol sustained-release capsules — allopurinol sustained-release capsules (0.25g), once a day, one pill at a time
  Arms: Treatment group
Drug: placebo capsules — placebo sustained-release capsules, once a day, one pill at a time
  Arms: Control group

SUMMARY:
The pathogenesis of coronary heart disease is closely related to inflammation. IL-1 beta is an effective target for anti-inflammatory treatment of coronary heart disease. Allopurinol is a drug used for treating hyperuricemia and gout for many years. Recently, allopurinol has been proved to inhibit the production of NLRP3 in monocytes and reduce the level of IL-1beta, resulting in the decrease of TNF-alpha, IL-6 and CRP. Thus, in this study, the investigators aim to evaluate the efficacy and safety of allopurinol sustained-release capsules on improving the stability of coronary plaque in patients with acute coronary syndrome treated by conventional standardized therapy by the single-center, prospective, randomized, double-blind and controlled methods, which would provide new strategies for the treatment of coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. the people who understand and would sign the informed consent voluntarily;
2. Aged 18 to 80 years old;
3. hospitalized patients diagnosed as acute coronary syndrome in the past 1 months;

   1. hsCRP > 2mg/L;
   2. allopurinol allergy gene HLA-B5801 was negative.

Exclusion Criteria:

1. history of coronary artery bypass grafting;
2. allergy to allopurinol or any excipient;
3. administration of allopurinol or other uric-acid-lowering drugs within 7 days before randomization;
4. abnormal liver function (ALT >1.5 fold of the upper limit);
5. renal dysfunction (creatinine clearance rate <45 ml/min);
6. thrombocytopenia (PLT<100g/L);
7. gout patients;
8. uncontrolled infectious diseases in screening period;
9. Thyroid dysfunction, moderate to severe anemia (hemoglobin < 90g/L), systemic lupus erythematosus, malignant hematopathy, leukopenia, asthma, inflammatory bowel disease and other immune diseases were found during the screening period;
10. Non-steroidal anti-inflammatory drugs, steroid hormone, immunomodulatory and chemotherapeutic drugs not included in the study protocol should be taken for a long time during the study period;
11. the history of surgery or interventional operation within 6 months before the screening period;
12. patients with mental disorders such as anxiety or depression;
13. pregnant women, lactating women or women of childbearing age who did not use effective contraceptive measures ;
14. patients who participated in other clinical trials 3 months before the screening period;
15. the researchers judged that patients were not suitable for this clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
low attenuation plaque volume | 12 months
  Changes of low attenuation plaque volume measured by coronary CTA

SECONDARY OUTCOMES:
total plaque volume | 12 months
  Changes of total plaque volume measured by coronary CTA
restructure index | 12 months
  Changes of restructure index measured by coronary CTA
inflammatory factors hsCRP | 12 months
  Changes of inflammatory factors hsCRP in plasma
All-cause mortality | 12 months
  All-cause mortality
Readmission rate of acute coronary syndrome | 12 months
  Readmission rate of acute coronary syndrome

OTHER OUTCOMES:
Adverse events and serious adverse events | 12 months
  Adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Revman